CLINICAL TRIAL: NCT05297708
Title: Office, Home, and Ambulatory Blood Pressure Measurements in Pediatric Patients
Brief Title: Office, Home, and Ambulatory Blood Pressure
Acronym: HBPA
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0843
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Elevated Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All Participants: he population would be pediatric patients 6 years to <19 years of age who were referred for elevated blood pressure. At the initial clinic visit, the participant will be consented and a thorough history will be taken. An ECHO and non-invasive vascular measurements will be taken (central BP, augmentation index, pulse wave velocity). Patients will have an ambulatory blood pressure monitor (ABPM) placed and be trained to use a home blood pressure monitor (HBP) which will be sent home with them. The monitors in this study are FDA-approved and are being used as indicated. After one day at home, patients will return the ABPM via mail and continue to take measurements with the HBP for 20 days.

SUMMARY:
This will be a prospective observational study. The population would be pediatric patients 6 years to <19 years of age who were referred for elevated blood pressure to investigate if home blood pressure (HBP) can determine blood pressure phenotype (normotensive, hypertensive, masked hypertension, white coat hypertension) as accurately as ambulatory blood pressure monitor (ABPM) in childhood and adolescence.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6 years to <19 years old;
2. Elevated blood pressure defined as 15% lower than the 95%ile BP based on clinical practice guidelines(CPG) but less than stage II hypertension based on CPG;
3. Tolerate ABPM 24 hours;
4. Tolerate HBP; and
5. Can have diabetes mellitus, obstructive sleep apnea, and attention deficit hyperactivity disorder managed by medication.
6. On stable doses of medications known to affect BP such as:

   1. Corticosteroids
   2. Calcineurin inhibitors
   3. Oral decongestants;
7. Clinically stable

Exclusion Criteria:

1. On antihypertension medications or treated in the last 6 months;
2. Pregnant;
3. Structural heart disease such as:

   1. Obstructive valvular disease
   2. Coarctation of the aorta
   3. Cardiomyopathy;
4. Other secondary causes such as:

   1. Renal artery stenosis
   2. Neurological condition with dysautonomia;
5. Recent initiation of medications known to affect BP such as:

   1. Corticosteroids
   2. Calcineurin inhibitors
   3. Oral decongestants;

Ages: 6 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: The population will be pediatric patients 6 years to <19 years years of age who were referred for elevated blood pressure to the Recruitment Hypertension clinic, Lipid Clinic, or Center for Better Health and Nutrition.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Determine blood pressure phenotype | 6-12 months after enrollment
  The primary objective of this study is to investigate if home blood pressure (HBP) can determine blood pressure phenotype (normotensive, hypertensive, masked hypertension, white coat hypertension) as accurately as ambulatory blood pressure monitor (ABPM) in childhood and adolescence.

SECONDARY OUTCOMES:
HBP correlation with end organ damage | 6-12 months after enrollment
  Our secondary objective is to determine if HBP correlates with end organ damage (i.e. elevated left ventricular mass, increased arterial stiffness, and decreased left ventricular strain) better than office BP. Our central hypothesis is that home blood pressure will accurately identify blood pressure phenotype and will correlate with end organ damage.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Urbina, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided